CLINICAL TRIAL: NCT05548855
Title: A Retrospective, Multicenter, International Study to Characterize the Natural History of Danon Disease
Brief Title: Natural History of Danon Disease
Status: Completed | Type: Observational
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-NI-A501-0122
Record Dates: First submitted 2022-07-29; First posted 2022-09-22 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-10

CONDITIONS: Danon Disease
Keywords: Danon Disease; Observational
MeSH Terms: conditions — Glycogen Storage Disease Type IIb | interventions — Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Transplant or Cardiac Assist Device: Female and male patients with confirmed diagnosis of Danon disease based on a genetic test positive for a mutation in LAMP2 For living patients who underwent heart transplantation or placement of a cardiac assist device, and for deceased patients, at least 1 MRI or echo assessment prior to heart transplantation/cardiac assist device placement or death.
  Interventions: Procedure: Heart Transplant; Device: Cardiac Assistive Device
- No Intervention: Female and male patients with confirmed diagnosis of Danon disease based on a genetic test positive for a mutation in LAMP2 for living patients (who have not undergone heart transplantation or placement of a cardiac assist device), availability of at least 6-month cardiology follow-up data

INTERVENTIONS:
Procedure: Heart Transplant — Patients who have undergone a heart transplant as standard of care (SOC) procedure
  Groups: Heart Transplant or Cardiac Assist Device
Device: Cardiac Assistive Device — Patients who have undergone a placement of a cardiac assistive device
  Groups: Heart Transplant or Cardiac Assist Device

SUMMARY:
This is a multicenter, international, non-interventional, natural history study designed to collect longitudinal retrospective clinical information on patients with Danon disease (DD). This study is composed of 2 parts:

* Feasibility study: to identify participating sites, assess site and team capabilities, confirm the site and investigator qualification for taking part in the study,
* Retrospective chart review: Data will be collected retrospectively by means of a chart review of living and/or deceased DD patients with a confirmed lysosome associated membrane protein-2 gene (LAMP2) mutation, and,
* For living patients (who have not undergone heart transplantation or placement of a cardiac assist device), availability of at least 6-month cardiology follow-up data,
* For living patients who underwent heart transplantation or placement of a cardiac assist device, and for deceased patients, at least 1 MRI or echo assessment prior to heart transplantation/cardiac assist device placement or death.

DETAILED DESCRIPTION:
Danon disease (DD) is a rare X-linked dominant genetic disorder characterized by cardiomyopathy, skeletal myopathy, and neurocognitive deficits. The disease is caused by a mutation in the lysosome associated membrane protein-2 gene (LAMP2). LAMP2 functions as a lysosomal membrane receptor in autophagy. Most men and many women with LAMP2 gene mutations will develop cardiac disease that includes hypertrophic cardiomyopathy and/or dilated cardiomyopathy, cardiac pre-excitation syndrome, and a propensity for arrhythmias. The prognosis is directly related to the severity of the cardiac disease, and many patients will die from sudden cardiac death. Males are typically more severely affected than females.

There is currently no therapy available to cure, or even prevent disease progression. DD treatment is thus primarily supportive therapy, and survival beyond 25 years without a cardiac transplantation is improbable for afflicted male patients.

Rocket Pharmaceuticals, a clinical-stage company advancing an integrated and sustainable pipeline of genetic therapies for rare pediatric disorders, is developing Rocket Pharmaceuticals Adeno-associated- vector-501 (RP-A501) (AAV9.LAMP2B), an investigational gene therapy product for DD and the first potential gene therapy for monogenic heart failure.

This retrospective, multicenter, international, longitudinal, non- interventional study of DD patients with confirmed LAMP2 mutation aims at characterizing the Natural History of disease in males and females. The Real-world data collected from patients in this natural history study will help support the overall development and protocol design of the RP-A501 gene therapy pivotal trial to be submitted to the health authorities.

Additionally, this study will allow identification of the core centers managing DD patients in several countries as well as the description of the disease characteristics, diagnosis pathway and disease progression. This will inform the development of patient profiles for future studies, including a potential prospective observational study to investigate the burden of disease among DD patients and an international patient registry for Danon disease.

The overarching goal of this retrospective, multicenter, international study is to gain a better understanding of the Natural History of Danon disease, by collecting de-identified information from patients with this condition treated.

Primary objective: Determine how specific cardiac manifestations in patients diagnosed with Danon disease change over time. Essential echocardiography and/or MRI-based parameters include: thickness of the Left Ventricular Posterior Wall at end-diastole (LVPWd); thickness of the Interventricular Septum at end-diastole (IVSd); Left Ventricular mass (LVmass); Left Ventricular Ejection Fraction (LVEF).

Secondary objectives: Describe the progression of other cardiac and extracardiac manifestations in patients diagnosed with Danon disease, including, but not limited to: serologic markers of heart failure, serologic markers of muscle injury, risk and frequency of arrhythmias, comprehensive echocardiogram and MRI-based assessments of cardiomyopathy, overall survival, and event-free survival (as defined subsequently).

Exploratory objectives:

1. Describe the diagnostic pathway of Danon disease, therapeutic management and local centers' approaches to genetic testing for LAMP2 mutations.
2. Identify key Natural History trends to inform a prospective European Union (EU) natural history study and plan for a potential gene therapy trial for DD patients in the EU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 6 years old and any sex.
2. Patients with a confirmed genetic mutation in LAMP2. 3a. Living patients (who have not undergone heart transplantation or placement of a cardiac assist device):

   * A minimum of 6 months of longitudinal data, including at least 2 echocardiograms or MRIs at least 6 months apart, prior to most recent follow-up visit or enrollment in Sponsor's gene therapy clinical trial.

     3b. Deceased patients or living patients who underwent heart transplantation or cardiac assist device placement:
   * At least 1 echocardiogram or MRI assessment prior to heart transplantation/ cardiac assist device placement or death

4. Informed consent/assent by the patient and/or their legally authorized representative (if the patient is living at the time of enrollment).

Exclusion Criteria:

1. Diagnosis of Danon disease without genetic testing confirmation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients with confirmed diagnosis of Danon disease based on a genetic test positive for a mutation in LAMP2
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Cardiac Manifestations- LVPWd | Retrospective minimum of 6 months
  Descriptive analysis will be conducted to characterize specific cardiac manifestations in patients diagnosed with Danon disease, and changes over time. Data collected will be analyzed by 6-month intervals and by the changes from initial evaluation over each 6-month interval. This includes the following cardiac parameters obtained from echocardiogram and/or MRI assessments: thickness of the left ventricular posterior wall end diastole and end systole (LVPWd).
Cardiac Manifestations- lVSd | Retrospective minimum of 6 months
  Descriptive analysis will be conducted to characterize specific cardiac manifestations in patients diagnosed with Danon disease, and changes over time. Data collected will be analyzed by 6-month intervals and by the changes from initial evaluation over each 6-month interval. This includes the following cardiac parameters obtained from echocardiogram and/or MRI assessments including thickness of the left ventricular systolic dysfunction (IVSd).
Cardiac Manifestations- LVmass | Retrospective minimum of 6 months
  Descriptive analysis will be conducted to characterize specific cardiac manifestations in patients diagnosed with Danon disease, and changes over time. Data collected will be analyzed by 6-month intervals and by the changes from initial evaluation over each 6-month interval. This includes the following cardiac parameters obtained from echocardiogram and/or MRI assessments including left ventricular mass (LVmass).
Cardiac Manifestations - LVEF | Retrospective minimum of 6 months
  Descriptive analysis will be conducted to characterize specific cardiac manifestations in patients diagnosed with Danon disease, and changes over time. Data collected will be analyzed by 6-month intervals and by the changes from initial evaluation over each 6-month interval. This includes the following cardiac parameters obtained from echocardiogram and/or MRI assessments including left ventricular ejection fraction (LVEF).

SECONDARY OUTCOMES:
Serologic Markers & Imaging - BNP | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of heart failure which include B-type natriuretic peptide (BNP).
Serologic Markers & Imaging Pro-BNP | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of heart failure which include Pro- B-type natriuretic peptide (Pro-BNP).
Serologic Markers & Imaging- CK-MB | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of heart failure which include creatine kinase - MB (CK-MB).
Serologic Markers & Imaging- Troponin | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of heart failure which include Troponin
Serologic Markers & Imaging- CPK | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of muscle injury, which include creatine phosphokinase (CPK).
Serologic Markers & Imaging- transaminases | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for serologic markers of muscle injury, which include transaminases
Serologic Markers & Imaging- Echo/MRI | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for the echocardiogram- and MRI-based assessments of cardiomyopathy, which include measures of cardiac hypertrophy or dilation
Serologic Markers & Imaging- BP | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for the echocardiogram- and MRI-based assessments of cardiomyopathy, which include measures of systolic and diastolic function
Serologic Markers & Imaging- GLS | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for the echocardiogram- and MRI-based assessments of cardiomyopathy, which include measures of Global Longitudinal Strain (GLS)
Serologic Markers & Imaging- E/A | Retrospective minimum of 6 months
  Mean values, standard deviations, medians and changes in means will be provided for the echocardiogram- and MRI-based assessments of cardiomyopathy, which include measures of mitral inflow ratio of the early (E) to late (A) (ventricular filling velocities (E/A))
Arrhythmias | Retrospective minimum of 6 months
  Time to event (risk of arrhythmia), for each of the following: supraventricular arrhythmias and non-sustained ventricular arrhythmias on Holter or similar monitoring, treatment with anti-arrhythmic medications
Wolf-Parkinson-White syndrome | Retrospective minimum of 6 months
  Time to event of Wolf-Parkinson-White syndrome (WPW) on electrocardiogram
ICD Placement | Retrospective minimum of 6 months
  Time to event of Implantable cardioverter-defibrillators (ICD) placement
Reason for ICD Placement | Retrospective minimum of 6 months
  Reasoning for ICD placement will be summarized by frequency of the reasons
Overall Survival | Retrospective minimum of 6 months
  Overall survival will be analyzed using Kaplan-Meier estimates. Patients lost to follow-up or who complete the study will be censored at the last follow-up time.
Event-free survival | Retrospective minimum of 6 months
  Event-free survival (EFS) will be analyzed using Kaplan-Meier estimates. EFS will be provided for Tier 1 events, Tier 1 + Tier 2 events, and Tier 1 + Tier 2 +Tier 3 events. Patients lost to follow-up or who complete the study will be censored at the last follow-up time.

CONTACTS AND LOCATIONS:
Locations (15):
- Institut klinické a experimentální medicíny (IKEM)- Institute for Clinical and Experimental Medicine, Prague, Czechia
- France (3):
  - CHU de Nantes, Hôpital Laennec, Nantes
  - APHP, Hôpital de la Pitié Salppêtrière - Charles Foix, Paris
  - CHU de Rennes, Hôpital Pontchaïllou, Rennes
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (3):
  - Ospedale Papa Giovanni XXIII di Bergamo ASST Pap Giovanni XXIII Hospital, Bergamo
  - University of Florence Dept. of Experimental and Clinical Medicine, Florence
  - IRCCS Burlo Garogolo- Hospital Burlo Garofolo, Trieste
- Spain (7):
  - Hospital Clínic de Barcelona - Barnaclínic+, Barcelona
  - Hospital Universitario de Bellvitge- Bellvitge University Hospital, Barcelona
  - Hospital Universitario La Paz - La Paz University Hospital, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda Puerta de Hierro Majadahonda - University Hospital, Madrid
  - Hospital Universitario Virgen de la Victoria- Virgen de la Victoria University Hosptial, Málaga
  - Hospital Álvaro Cunqueiro, Pontevedra
  - Hospital Universitario y Politécnico La Fe, Instituto De Investigación Sanitaria La Fe, La Fe University and Polytechnic Hospital, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Glycogen Storage Disease type IX — https://medlineplus.gov/genetics/condition/glycogen-storage-disease-type-ix/
- See also: Danon Disease — https://medlineplus.gov/genetics/condition/danon-disease/
- See also: Danon Disease — https://rarediseases.info.nih.gov/diseases/9730/danon-disease